CLINICAL TRIAL: NCT05603481
Title: Glucose Monitoring in Patients With Eating Disorders: A Pilot Study
Brief Title: CGM in Patients With ED's
Acronym: CGM
Status: Completed | Type: Observational
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Principal Investigator, Kristin Sterrett, Kristin Sterrett, Hospitalist, Principal Investigator, Denver Health and Hospital Authority
Other Study IDs: DenverHealth
Record Dates: First submitted 2022-07-29; First posted 2022-11-02 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Anorexia Nervosa Restricting Type; Anorexia Nervosa, Binge Eating/Purging Type; ARFID; Avoidant Restrictive Food Intake Disorder
Keywords: CGM; Continuous Glucose Monitor; ACUTE
MeSH Terms: conditions — Anorexia Nervosa; Bulimia; Avoidant Restrictive Food Intake Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- CGM
  Interventions: Device: Continuous Glucose Monitor

INTERVENTIONS:
Device: Continuous Glucose Monitor — Patients will wear a CGM device on their arm for 10 days, while receiving standard of care blood draws and finger stick sugar checks.

SUMMARY:
To determine the accuracy of continuous glucose monitoring (CGM) with point of care (POC) fingerstick glucose monitoring and venous blood glucose in patients with eating disorders, specifically anorexia nervosa, restricting subtype (AN-R); avoidant/restrictive food intake disorder (ARFID); and anorexia nervosa, binge/purge subtype (AN-BP).

DETAILED DESCRIPTION:
It is the experience of the treatment team at ACUTE Center for Eating Disorders and Severe Malnutrition that POC fingerstick testing can be inaccurate in patients when POC fingerstick testing is compared to serum glucose values. However, this has not been formally studied.

This study seeks to define the accuracy of POC fingerstick testing and CGM as compared to blood serum glucose monitoring via phlebotomy. It also seeks to better understand the frequency of hypo- and hyperglycemia in this population using continuous glucose monitoring during the first 10 days of admission. Ideally, an accurate method of monitoring glucose values in this population beside phlebotomy draws needs to be established.

Blood will be drawn shortly after participants admission to the unit as part of usual care and will continue to be drawn daily as usual care for the next 5 days. Patient blood sugar will be checked daily using POC finger sticks until hypoglycemia resolves. If patient choose to participate in this study, the investigators will do additional POC testing on days 6 and 8 POC finger sticks will be done 30-minutes post breakfast/lunch/dinner. On the same day the patient agrees to be in this study, the patient will have a Dexcom CGM placed to the back of their arm, or on another area of the body depending on the recommendation from the manufacturer (DEXCOM). Patient will wear the CGM for the full 10 days that the study is being conducted.

Patient will also be asked to complete a simple log regarding the date and time the patient received post Breakfast/lunch/dinner POC tests on days 6 and 8. The patient may ask the PSCA Patient Safety Care Attendant (PSCA) to assist patient with this task.

Data received from the Dexcom device will automatically be uploaded to the Dexcom cloud. Only the research statistician will have access to these data. Staff from Dexcom do not have access to these data.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65 and meet the DSM-V criteria for AN-R or AN-BP or ARFID
* Admission %IBW ≤ 75%

Exclusion Criteria:

* Diagnosed with an eating disorder other than AN-R or AN-BP or ARFID
* %IBW > 75% on admission
* Inability to give informed consent to participate/lacks decisional capacity
* Unable to follow the study protocol
* Transferred to the unit on a mental health hold/short term certification
* Treatment team refusal of patient's participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seeking care for medically compromised severe eating-disorders. Weight less than 75% of the patient's ideal body weight (IBW). a history of serious medical complications related to the eating disorder (electrolyte imbalance, fluid problems, organ failure, cardiac irregularities or gastrointestinal complications); a need to detoxify from, or avoid complications from, a purging behavior (vomiting, laxative or diuretic abuse); and/or need for additional medical workup/oversight to determine if a presenting problem is psychiatric or medical in nature.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Determine the accuracy of continuous glucose monitors (CGM) | 10 days
  To perform statical analysis to verify the accuracy of interstitial glucose measured via CGM as compared to the POC finger stick. In individuals with severe malnutrition, secondary to eating disorders
Serum glucose fluctuations | 10 days
  To better understand changes in serum glucose as a function of fasting and nutritional completion as measured via interstitial glucose values as reported by the CGM.
Frequency of hypoglycemia | 10 days
  To better understand the frequency of hypoglycemia measured via interstitial glucose values as reported by the CGM.

SECONDARY OUTCOMES:
Difference in glucose levels | 10 days
  To statically analyze the similarities and differences of interstitial glucose monitoring using CGM amongst patients with AN-R vs AN-BP vs ARFID.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Sterrett, MD, Principal Investigator — Denver Health and Hospital Authority
Locations (1):
- Denver Health and Hospital Authority, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No